CLINICAL TRIAL: NCT03383198
Title: Pectoralis (II) Block With Liposomal Bupivacaine vs Bupivacaine Plus Dexamethasone for Mastectomy With Immediate Reconstruction
Brief Title: Pectoralis (II) Block With Liposomal Bupivacaine vs Bupivacaine for Breast Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Early termination due to manufacturer discontinued supplying the product for the study.
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00072519
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2018-08

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Only anesthesiologist performing injection will be aware of which side is injected with each drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liposomal Bupivacaine Left (Active Comparator): Liposomal Bupivacaine left injection. Liposomal Bupivacaine is injected on the left, Bupivacaine plus Dexamethasone on the right
  Interventions: Drug: Liposomal bupivacaine left injection
- Liposomal Bupivacaine Right (Active Comparator): Liposomal Bupivacaine right injection. Liposomal Bupivacaine injected on the right, Bupivacaine plus Dexamethasone on the left
  Interventions: Drug: Liposomal bupivacaine right injection

INTERVENTIONS:
Drug: Liposomal bupivacaine right injection — Right side will have liposomal bupivacaine ultrasound guided PEC II field block injection ; the left side side will have bupivacaine plus dexamethasone ultrasound guided PEC II field block injection.
  Other Names: Exparel Right
  Arms: Liposomal Bupivacaine Right
Drug: Liposomal bupivacaine left injection — Left side will have liposomal bupivacaine ultrasound guided PEC II field block injection ; the right side side will have bupivacaine plus dexamethasone ultrasound guided PEC II field block injection.
  Other Names: Exparel Left
  Arms: Liposomal Bupivacaine Left

SUMMARY:
This is a randomized controlled pilot study evaluating length of pain control with either liposomal bupivacaine or with bupivacaine plus decadron after PEC II injection in patients having bilateral mastectomies with immediate reconstruction.

DETAILED DESCRIPTION:
This research hopes to determine the duration of patient-reported analgesia provided by ultrasound guided PEC II field block injections. The design of the study randomly assigns the side of injection of the study drugs into each patient. All patients are having bilateral mastectomy with immediate reconstruction. Visual analog pain scores (VAS) will be recorded serially for both sides of the patient's chest in hopes of determining a difference in duration and efficacy of the two drugs. In addition to VAS scores, a subjective, binary question will be our primary outcome: does one side of your chest have more surgical pain than the other? We hope that his question, despite being entirely subjective, overcomes interpatient variability of numerical pain score reporting.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for bilateral mastectomy

Exclusion Criteria:

* allergy to local anesthetics, prior breast surgery, asymmetric surgical plan

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Bilateral mastectomy
Enrollment: 5 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Hand, MD, Principal Investigator — Prisma Health-Upstate
Locations (1):
- Patewood Memorial Hospital, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bashandy GM, Abbas DN. Pectoral nerves I and II blocks in multimodal analgesia for breast cancer surgery: a randomized clinical trial. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):68-74. doi: 10.1097/AAP.0000000000000163. PMID 25376971
- [Background] Amundson AW, Johnson RL, Abdel MP, Mantilla CB, Panchamia JK, Taunton MJ, Kralovec ME, Hebl JR, Schroeder DR, Pagnano MW, Kopp SL. A Three-arm Randomized Clinical Trial Comparing Continuous Femoral Plus Single-injection Sciatic Peripheral Nerve Blocks versus Periarticular Injection with Ropivacaine or Liposomal Bupivacaine for Patients Undergoing Total Knee Arthroplasty. Anesthesiology. 2017 Jun;126(6):1139-1150. doi: 10.1097/ALN.0000000000001586. PMID 28234636

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liposomal Bupivacaine Left | Liposomal Bupivacaine Right
Started | 4 | 1
Completed | 4 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients undergoing bilateral mastectomy with immediate reconstruction at Greenville Memorial Hospital or Patewood Memorial Hospital.
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine Left | Liposomal Bupivacaine Right | Total
Number analyzed (Participants) | 4 | 1 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 59.25 [48 to 71] | 44 [44 to 44] | 56.2 [44 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 1 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Subjective Bilateral Pain Comparison
Description: Subjective, binary question "Does one side of your chest have more surgical pain than the other?"
Time Frame: up to 48 hours
Population: Patients undergoing bilateral mastectomy with immediate reconstruction by breast surgeons at Greenville Health System.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine Left | Liposomal Bupivacaine Right
Number analyzed (Participants) | 4 | 1
Participants | 1 | 0

2. Secondary Outcome: Duration of Analgesia
Description: Duration of analgesia perception by patient measured bilaterally using Visual Analog Scale
Time Frame: up to 48 hours
Population: Patients undergoing bilateral mastectomy with immediate reconstruction by breast surgeons at Greenville Health System.
Measure: Mean (Full Range); unit: hours
Arm/Group | Liposomal Bupivacaine Left | Liposomal Bupivacaine Right
Number analyzed (Participants) | 4 | 1
hours | 21.5 [8 to 42] | 36 [36 to 36]

ADVERSE EVENTS:
Time Frame: 48 hours
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information does not differ from the clinicaltrials.gov definitions.
Groups:
- Liposomal Bupivacaine: Liposomal Bupivacaine left injection. Liposomal Bupivacaine is injected on the left, Bupivacaine plus Dexamethasone on the right
  Liposomal bupivacaine left injection: Left side will have liposomal bupivacaine ultrasound guided PEC II field block injection ; the right side side will have bupivacaine plus dexamethasone ultrasound guided PEC II field block injection.
- Bupivacaine Plus Dexamethasone: Liposomal Bupivacaine right injection. Liposomal Bupivacaine injected on the right, Bupivacaine plus Dexamethasone on the left
  Liposomal bupivacaine right injection: Right side will have liposomal bupivacaine ultrasound guided PEC II field block injection ; the left side side will have bupivacaine plus dexamethasone ultrasound guided PEC II field block injection.
Arm/Group | Liposomal Bupivacaine | Bupivacaine Plus Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. Manufacturer discontinued supplying product for the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT03383198/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT03383198/ICF_001.pdf